CLINICAL TRIAL: NCT04954014
Title: Pilot Study of Single Dose Bevacizumab as Treatment for Acute Respiratory Distress Syndrome (ARDS) in COVID-19 Patients
Acronym: BEVACOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of financing, lack of COVID19 patients in the ICU.
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEVACOR
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: ARDS, Human; Coronavirus Infection
Keywords: ARDS; SARS-CoV-2; Bevacizumab
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Phase II, multi-centered, randomized, open label, two-armed clinical trial to study the safety and efficacy of bevacizumab in COVID-19 positive patients who consequently developed ARDS (acute respiratory distress syndrome) and who have previously received anti-viral and anti-inflammatory treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEVACIZUMAB (Experimental): Patients will receive best available treatment (BAT) for COVID-19 plus single dose bevacizumab calculated as 7,5 mg/kg diluted in 250cc of saline solution during 90 minutes.
  Interventions: Drug: Bevacizumab
- BEST AVAILABLE TREATMENT (Active Comparator): Patients will receive best available treatment for COVID-19.
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive best available treatment (BAT) for COVID-19 plus a single dose of bevacizumab calculated as 7,5 mg/kg diluted in 250cc of saline solution during 90 minutes.
  Arms: BEVACIZUMAB
Drug: BAT — Patients will receive best available treatment for COVID-19.
  Arms: BEST AVAILABLE TREATMENT

SUMMARY:
Our hypothesis is that treating ARDS caused by COVID-19 with bevacizumab improves mortality. This is a phase II, multi-centered, randomized, open label, two-armed clinical trial to study the safety and efficacy of bevacizumab in COVID-19 positive patients who consequently developed ARDS (acute respiratory distress syndrome) and who have previously received anti-viral and anti-inflammatory treatment.

DETAILED DESCRIPTION:
The vascular endothelial growth factor (VEGF) improves vascular capillarity, which plays an important role in the uncontrolled inflammatory reaction that happens in ARDS. As opposed to this event, angiogenic therapy (like bevacizumab) is known to contribute to normal vascularization, relevant for regaining vascular permeability. Studies in animal models have shown that treating ARDS with anti-VEGF therapy is effective.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 and under 90 years old.
* Confirmed COVID-19 positive diagnostic through PCR.
* Radiological image compatible with non-cardiogenic bilateral pleuropulmonary exudate.
* Patient has received anti-viral and anti-inflammatory therapy.
* Present any of the following clinical-functional criteria:

  1. Respiratory distress: Tachypnea> 30 breaths / minute
  2. Partial arterial oxygen pressure (PaO2) / Fraction of inspiration (FiO2) ≤ 300 mmHg
* Signed informed consent, directly or delegated.

Exclusion Criteria:

* Severe liver dysfunction (Child Pugh ≥ 3 or AST> 5 times normal)
* Severe renal dysfunction with glomerular filtration <30 mL / minute or under treatment with hemodialysis or peritoneal dialysis.
* Poorly controlled hypertension (BPs> 160 mmHg or TAd <100 mmHg) or having a history previous hypertensive crisis or hypertensive encephalopathy.
* History of poorly controlled heart disease with a NYHA> 2.
* History of thrombosis in the previous 6 months.
* Signs of active bleeding.
* Open wounds, gastrointestinal perforation.
* Diagnosis of thrombophilic diseases or hemorrhagic diathesis.
* Active viral hepatitis or HIV not properly treated.
* Intolerance or allergy to bevacizumab or its components.
* Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | After 28 days
  Mortality

SECONDARY OUTCOMES:
PaO2/FiO2 | 6 hours before bevacizumab administration and 24 hours,72 hours,7 days,14 days and 28 days after.
  Ratio calculation
Clinical improvement according to scale recommended by WHO for COVID19 | 24 hours, 72 hours, 7 days, 14 days and 28 days after treatment.
  Clinical improvement according to WHO scale (World Health Organization) for COVID19 which goes from 1 to 7 points.
Time to clinical improvement as stated in the National Early Warning Score 2 (NEWS) | From randomization until improvement of 2 points in the scale or until hospital discharge, whatever happens first, assessed up to 28 days.
  NEWS assesses clinical risk on a scale of 1 (low) to 8 (high)
Time to improvement of oxygenation | From randomization until outcome event assessed up to 28 days.
  Improvement shown during, at least, 48 hours.
Time to improvement of Sp2/O2 ratio regarding the worst Sp2/O2 ratio obtained before bevacizumab treatment. | From randomization until first documented Sp2/O2 ratio improvement, assessed up to 28 days.
  Time to improvement of Sp2/O2 ratio regarding the worst Sp2/O2 ratio obtained before bevacizumab treatment
Time to absence of oxygen need to maintain a saturation equal or over 93% | From randomization until patient doesn't need oxygen to mantain 93% saturation, assessed up to 28 days.
  Time to absence of oxygen need to maintain a saturation equal or over 93%
Favorable radiological evaluation. | From randomization until first documented radiology improvement, assessed up to 28 days.
  Dictated by 3 radiologists.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: When study is published.
Access Criteria: Send request to access.